CLINICAL TRIAL: NCT06653764
Title: Effects of Chest Physiotherapy and Aerobic Exercise Training in Improving Physical Fitness InYoung Children Post Abdominal Surgery: an Experimental Trial
Brief Title: Chest Physiotherapy and Aerobic Training in Children Post Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Vandana Esht, Associate Professor, University of Jazan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: REF20241002
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Post Abdominal Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rehabilitation (Experimental)
  Interventions: Other: Chest physiotherapy and aerobic exercise training

INTERVENTIONS:
Other: Chest physiotherapy and aerobic exercise training — Chest Physiotherapy including Percussion, vibration and shaking; along with it aerobic exercises such as walking up and down stairs, bedside ambulation, step walking

SUMMARY:
This study will underscore the clinical importance of integrating chest physiotherapy and aerobic exercise training into the post-abdominal surgery care regimen for young children.By improving physical fitness levels, these interventions contribute significantly to the overall recovery process and enhance the well-being of pediatric patients. Implementing such strategies can optimize functional outcomes, reduce complications, and promote a faster return to normal activities, thereby improving the quality of life for young patients undergoing abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age from 5 Years to 15 Years, Gender: Both, Details: Children who underwent abdominal surgery, having stable vitals, admitted in PICU and pediatric wards

Exclusion Criteria:

* Patients with severe neurological illness, uncooperative patients, comatose patients, patients who are unwilling to enroll in study

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2024-07-10 (Actual); Primary Completion 2024-08-11 (Actual); Study Completion 2024-08-11 (Actual)

PRIMARY OUTCOMES:
Spirometey, manual muscle testing | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Arogyam Institute ofParamedical and AlliedSciences, Roorkee, Uttarakhand, India